CLINICAL TRIAL: NCT03285009
Title: Optimizing Body and Movement Specific Characteristics in Volleyball Players to Reduces Injuries in Young Athletes.
Brief Title: Movement Patterns in Young Volleyball Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, Prof. Dr. F. Staes, Professor, Head of Musculoskeletal Research Group, Universitaire Ziekenhuizen KU Leuven
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S60760
Record Dates: First submitted 2017-09-10; First posted 2017-09-15 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Injuries; Training; Athlete; Youth
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Masking Description: Masking not possible as individual treatment is given
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Training intervention (Other): See information elsewhere
  Interventions: Other: Training intervention

INTERVENTIONS:
Other: Training intervention — Based on the baseline screening, which is part of the normal prevention routine within the school, all athletes are given individual advice with regard to points of attention within training. For example: those athletes with reduced balance, will get more balance training.
  Intervention is individual as said and will be guided and supervised by the physical trainer and medical staff of the school.

SUMMARY:
This project is a consequence of the research chair project studying the same phenomenon in adult volleyball players. The project will make use of and be part of the routine medical screening that is taken by the young players of the first degree of the Leuven Volleyball School, Belgium. All young players must undergo a routine medical investigation and movement screening. This is obliged by the law. The current project will use these data. Outcome parameters will be used to advice the trainer staff of the school to adjust their training interventions. This is normal routine too as the involved medical department has been advising the school for many years. Players will be followed up for 6 weeks. After those 6 weeks, the movement screening will be repeated to evaluate the change in the different outcome parameters. This last screening is not part of a normal routine as players normally are investigated more in a subjective way. The medical team and school want to change that routine.

Data will be used to further improve training modalities and sports performance and reduce injury risk in these young athletes.

ELIGIBILITY:
Inclusion Criteria:

* All students from the first degree of the Volleyball school will participate
* Male and female athletes will be included
* Signing of an informed consent and assent form (for young kids) to use data for research
* Agreement given by the medical staff to use data and allowing the kids to be accepted by the school

Exclusion Criteria:

* When inclusion criteria are not met

Ages: 11 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2017-09-25 (Actual); Primary Completion 2018-12-23 (Actual); Study Completion 2018-12-23 (Actual)

PRIMARY OUTCOMES:
Change of joint mobility | Difference between baseline and 6 weeks
  Mobility will be assessed by using goniometer measurements (degrees of movement)
Change of strength | Difference between baseline and 6 weeks
  Strength will be assessed by using handheld dynamo-meter data (Newton)
Change in balance score | Difference between baseline and 6 weeks
  Stability is measured using the score on the Star Excursion Balance Test (numeric score on balance scale)
Change in lower limb joint angles during a single leg drop vertical jump | Difference between baseline and 6 weeks
  Movement quality is measured using joint angles (trunk, pelvis, hip, knee, ankle)
Change in lumbopelvic stability score | Difference between baseline and 6 weeks
  Lumbopelvic stability is scored using 9 clinical tests (Bend knee fall out, Active straight leg raise, prone knee bend, sitting knee extension, standing bow, pelvic tilt, one leg stance, backward rocking, forward rocking). Each test is given a score between 0 (poor performance) and 2 (good performance) adding up to a total score of 18.
Change in lower limb joint angles during a drop jump | Difference between baseline and 6 weeks
  Movement quality is measured using joint angles (trunk, pelvis, hip, knee, ankle)

SECONDARY OUTCOMES:
Individualized web diagram of all outcome measurements | Baseline
  Baseline data on joint mobility (joint angles), strength (N), balance (Star Excursion Balance Test Score, lumbopelvic control scores) and joint angles during a drop jump and single leg drop vertical jump) are all visualized on a web diagram per athlete
Number of injuries | Baseline information from medical investigation
  Description of number of injuries

CONTACTS AND LOCATIONS:
Overall Officials: Filip F Staes, prof, Principal Investigator — KU Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared with other researchers. Data will be available to the medical and trainers staff. For research purposes, all data will be made anonymous.